CLINICAL TRIAL: NCT01021566
Title: Advances in Opiate Detoxification Using the Combined Hemoperfusion-hemodialysis: A Comparison Study With Conventional Methadone Treatment (HPDMT)
Brief Title: Opiate Detoxification Using the Combined Hemoperfusion-hemodialysis
Acronym: HPDMT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First People's Hospital of Foshan (Other)
Responsible Party: the First People's Hospital of Foshan, the First People's Hospital of Foshan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 075783161516
Expanded Access: Available
Record Dates: First submitted 2009-11-27; First posted 2009-11-30 (Estimated); Last update posted 2009-11-30 (Estimated); Status verified 2009-11

CONDITIONS: Opiate Addiction
Keywords: Opiate addiction; Withdrawal symptoms; hemoperfusion; hemodialysis; methadone
MeSH Terms: conditions — Opioid-Related Disorders; Substance Withdrawal Syndrome | interventions — Methadone

ARMS (2):
- Combined hemoperfusion-hemodialysis (Experimental): On admission thirty patients will receive the combined hemoperfusion-hemodialysis treatment regimen three hours everyday for three days.
  Interventions: Device: Combined hemoperfusion-hemodialysis
- Methadone, conventional treatment for opiate detoxification (Active Comparator): On admission thirty patients receive the 10-day methadone treatment regimen.
  Interventions: Drug: Methadone

INTERVENTIONS:
Device: Combined hemoperfusion-hemodialysis — Combined hemoperfusion-hemodialysis for opiate detoxification for 3 days
  Arms: Combined hemoperfusion-hemodialysis
Drug: Methadone — On admission all patients will undergo a 3-day stabilization period. Then they will begin the 10-day methadone treatment regimen. The starting dose of methadone is determined by the mean daily dose requirement during the stabilization period and the dose will be reduced to zero at a linear rate over the 10 days treatment.
  Arms: Methadone, conventional treatment for opiate detoxification

SUMMARY:
The purpose of this study is to determine whether combined hemoperfusion-hemodialysis treatment is an alternative drug-free, effective, and safe treatment for opiate detoxification.

DETAILED DESCRIPTION:
Drug abuse remains a major society problem in our community and is also a major health problem in our modern society. Thus, education to prevent the young generation to avoid drug abuse and detoxification to help those to quite from the drug abuse are two major key steps in the controlling drug abuse program.

Currently, medications for opiate detoxification, such as methadone, are commonly used worldwide. However, methadone is also an addictive medication. When it is stopped suddenly, patients usually produce unpleasant withdrawal symptoms. Meanwhile, methadone is also potentially to be abused too. Thus, it is urgently needed to seek an alternative safer, effective, drug-free method for opiate detoxification. Based on our clinical observation, the timely clearance of toxicities from the body or blood is a safe and effective detoxification method. Thus, we hypothesized that the use of combined hemoperfusion-hemodialysis may be an alternative drug-free, effective, and safe treatment for opiate detoxification. This will be tested in patients who have severe drug abuse and are under custodial conditions by a daily combined hemoperfusion-hemodialysis for 3 days. The efficacy and safety of the hemoperfusion-hemodialysis will be compared to a 10 day standard methadone detoxification treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be fulfilled DSM-IV criteria(American Psychiatric Association) for opiate dependence.
* A history of current dependence on heroin, which was supported by laboratory results from urine drug screening, using both chromatographic and radioimmunoassay methods.
* Opioid dependent patients who inject heroin from 0.5g to 1.0g daily by veins for at least 1 year.
* Haven't received methadone treatment for at least 2 months before entry to this study.
* Be able to understand and have signed the informed consent.

Exclusion Criteria:

* Take heroin for the first time.
* Positive for HIV.
* The function of cruor or hemorrhage is badly damaged.
* The number of platelets is lower than 70×10*9.
* Co-dependent on substances other than opiates (including alcohol, benzodiazepines, cocaine, or amphetamines).
* Methadone dose requirement is over 70 mg/day as determined by the 3-day dose assessment period.
* Have serious physical illness or major psychiatric illness.
* Pregnant woman.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
The Short Opiate Withdrawal Scale(SOWS-Gossop) | 15 days

SECONDARY OUTCOMES:
Blood levels of morphine and β-endorphin, and the urine level of morphine. | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- the First People's Hospital of Foshan, Foshan, Guangdong, China